CLINICAL TRIAL: NCT02791659
Title: Radiation Exposure of ERCP Personnel at Different Standing Locations and Different Patient Positions (Prone and Left Lateral Decubitus)
Brief Title: Radiation Exposure of ERCP Personnel at Different Standing Locations and Different Patient Positions.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PA-E-RAD002
Record Dates: First submitted 2016-06-01; First posted 2016-06-07 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Occupational Radiation Exposure
Keywords: radiation exposure; ERCP; prone; left lateral decubitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Left lateral decubitus (Active Comparator): In this group, the position will be assigned to Left lateral decubitus during ERCP. The radiation from fluoroscopy will be adjusted by automatic beam adjustment function to obtain the image quality.
  Interventions: Radiation: Automatic beam adjustment function
- Prone (Experimental): In this group, the position will be assigned to Prone during ERCP. The radiation from fluoroscopy will be adjusted by automatic beam adjustment function to obtain the image quality.
  Interventions: Radiation: Automatic beam adjustment function

INTERVENTIONS:
Radiation: Automatic beam adjustment function — The fluoroscopy system has an automatic beam adjustment function to maintain a good quality of image output.

SUMMARY:
X-ray beam produced during endoscopic retrograde cholangiopancreatography (ERCP) affect not only the patient, but the personnel of ERCP team may have the effect from the scattered ray. According to the automatic beam adjustment function, the thicker object (eg. lying left lateral) might produce higher scatter ray than thinner object (eg. lying prone). The investigators evaluate the radiation exposure among ERCP personnel compare between patient's 2 different positions.

DETAILED DESCRIPTION:
Personal solid-state dosimeters were used to measure the radiation dose on personnel during ERCP procedure. The real-time effective doses were displayed at a monitoring screen. A dosimeter was attached outside thyroid collar of each ERCP team member included of 1st endoscopist, 2nd endoscopist, and nurse anesthetist.

Patients' age, gender, BMI, body thickness, and indications for ERCP were recorded. The patients were randomized into 2 groups by block-of-four. The patients' position was assigned to prone or left lateral decubitus. Each ERCP personnel wore a lead apron and the dosimeter was attached outside the thyroid collar. The ERCP procedure was performed according to the indication in a standard technique. After ERCP procedure, the total fluoroscopic time (minute), fluoroscopy tube voltage (kV), fluoroscopy tube current (mA), patient entrance skin dose (mGy) and personnel effective dose (Sv) from each dosimeter were recorded.

Continuous variables were compared by Student's t-test or Man Whitney U-test, where appropriate. Categorical variables were compared by Chi-square or the Fisher exact test. Statistical analysis was calculated by using SPSS statistical software (version17 for Window, Chicago, USA) and two sided p-value < 0.05 was considered to be statistical significant.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for ERCP

Exclusion Criteria:

* pregnancy
* American Society of Anesthesiologists (ASA) physical status class III - IV
* unstable vital signs
* patients' position needed to be changed during the procedure
* patients who need fixed position for ERCP (such as biliary hilar lesion)
* enteroscope-assisted ERCP
* the consent form can not be obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rungsun Rerknimitr, MD, FRCP, Principal Investigator — Chulalongkorn University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Left Lateral Decubitus | Prone
Started | 27 | 28
Completed | 27 | 27
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Left Lateral Decubitus | Prone | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [51 to 76.5] | 67 [59 to 73] | 67 [55.25 to 75.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 10 | 15 | 25
BMI [Mean (Standard Deviation); unit: kg/m2] | 22.9 (3.45) | 22.2 (4.07) | 22.5 (3.77)
Indication for ERCP [Count of Participants; unit: Participants]
  Choledocholithiasis | 18 | 17 | 35
  Malignant biliary obstruction | 6 | 8 | 14
  Benign biliary obstruction | 3 | 2 | 5
Vertical thickness [Mean (Standard Deviation); unit: cm] | 27.2 (3.71) | 20.2 (4.18) | 23.7 (5.31)
Fluoroscopy time [Median (Inter-Quartile Range); unit: min] | 4.06 [2.58 to 6.10] | 4.14 [2.76 to 5.82] | 4.11 [2.58 to 6.03]
Dose area product [Median (Inter-Quartile Range); unit: Gy-cm2] | 22.3 [17.55 to 40.15] | 23.2 [16.25 to 32.10] | 22.65 [16.75 to 37.2]
Patient entrance skin dose [Mean (Inter-Quartile Range); unit: mGy/min] | 5.7 [4.76 to 7.56] | 5.5 [4.88 to 5.89] | 5.6 [4.86 to 6.72]

OUTCOME MEASURES:

1. Primary Outcome: Effective Radiation Dose
Description: The effective radiation which represents equivalent dose to eye lens of each personnel were compared between 2 groups.
Time Frame: Immediate after procedure
Measure: Median (Inter-Quartile Range); unit: mSv
Arm/Group | Left Lateral Decubitus | Prone
Number analyzed (Participants) | 27 | 27
mSv | 0.0307 [0.0192 to 0.0437] | 0.0192 [0.0115 to 0.0322]

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Left Lateral Decubitus | Prone
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes